CLINICAL TRIAL: NCT02741830
Title: Long Term Outcomes of Uterosacral Ligament Suspension Versus Robotic Sacrocolpopexy
Brief Title: Uterosacral Ligament Suspension vs Robotic Sacrocolpopexy
Status: Completed | Type: Observational
Sponsor: TriHealth Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: 16-003
Record Dates: First submitted 2016-04-13; First posted 2016-04-18 (Estimated); Last update posted 2019-01-10 (Actual); Status verified 2018-02

CONDITIONS: Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Uterosacral ligament suspension (USLS): This group of patients underwent the procedure of native tissue vaginal reconstructive surgery using uterosacral ligament suspension for pelvic organ prolapse.
- Robotic sacrocolpopexy (RSC): This group of patients underwent the reconstructive pelvic surgery of robotic sacrocolpopexy using synthetic mesh.

SUMMARY:
This cross sectional, two cohort study seeks to investigate both anatomic outcome and subjective, functional outcome of uterosacral ligament suspension versus robotic sacrocolpopexy and compare patient satisfaction, bladder function, sexual function and complication rate for each procedure.This study will provide a better understanding about the durability of these procedures and long term complication.

DETAILED DESCRIPTION:
Pelvic organ prolapse is a common problem affecting many women and there is a 12.6% lifetime risk of undergoing reconstructive pelvic surgery. There are several surgical options available to patients undergoing reconstruction for pelvic organ prolapse, however addressing the apex is recommended to achieve the most durable outcomes. Two of the most commonly performed procedures for apical prolapse repair are uterosacral ligament suspension and robotic sacrocolpopexy.

High uterosacral ligament suspension is a native tissue repair which is performed by affixing the vaginal apex to the bilateral uterosacral ligaments using permanent or delayed-absorbable sutures. This is performed typically in a vaginal approach. Sacrocolpopexy is a performed by attaching the anterior and posterior vaginal walls to the sacral promontory using synthetic mesh, typically polypropylene. This procedure can be performed by an abdominal approach, a laparoscopic approach or with the assistance of the da Vinci robotic system. In recent years, robotic sacrocolpopexy has largely replaced the abdominal approach, and become the procedure of choice for minimally invasive surgeons.

Most studies evaluating sacrocolpopexy outcomes were performed prior to the popularity of robotics and therefore concentrate on abdominal sacrocolpopexy.

This cross sectional, two cohort study will compare outcomes of uterosacral ligament suspension versus robotic sacrocolpopexy and will give pelvic surgeons a better understanding about the durability of these procedures, and possible longer term complication rates.

Subjects will be contacted and asked to come to the office for a visit and completion of questionnaires. If they cannot come to the office, an Informed Consent Form (ICF) and questionnaires will be mailed to them to complete and return separately.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 years of age or older who spent 3-7 years following uterosacral ligament suspension or robotic sacrocolpopexy.
* Concurrent procedures such as suburethral sling, bilateral salpingoophorectomy, hysterectomy, rectopexy.
* Concurrent procedures such a s takedown of sling

Exclusion Criteria:

* Concurrent procedure to remove vaginal mesh at time of their index surgery
* Unwillingness to participate in the study
* Dementia or inability to provide informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All women 18 years of age or older who underwent the uterosacral ligament suspension or robotic sacrocolpopexy for treatment of pelvic organ prolapse 3-7 years ago.
Sampling Method: Non-Probability Sample
Enrollment: 186 (Actual)
Dates: Start 2016-04-07 (Actual); Primary Completion 2018-05-21 (Actual); Study Completion 2018-10-16 (Actual)

PRIMARY OUTCOMES:
Subject patient symptoms of prolapse, "bulge" symptom | 3-7 years after reconstructive surgery involving uterosacral ligament suspension or robotic sacrocolpopexy
  This is a binary outcome, and success is defined as answering "No" to question #3 on the Pelvic Organ Prolapse Distress Inventory (PFDI-20) questionnaire, as well as the absence of any reoperation or pessary use for pelvic organ prolapsed.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Pauls, MD, Principal Investigator — TriHealth - Cincinnati Urogynecology Associates
Locations (1):
- Cincinnati Urogynecology Associates, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Smith BC, Crisp CC, Kleeman SD, Yook E, Pauls RN. Uterosacral Ligament Suspension Versus Robotic Sacrocolpopexy for Treatment of Apical Pelvic Organ Prolapse. Female Pelvic Med Reconstr Surg. 2019 Mar/Apr;25(2):93-98. doi: 10.1097/SPV.0000000000000704. PMID 30807407